CLINICAL TRIAL: NCT00277602
Title: A Phase III Multicenter, Double-Blind, Parallel-Group, Placebo Controlled Study to Measure the Effect of Riluzole 50 mg b.i.d. Over a Period of Three Years on the Progression of Huntington's Disease
Brief Title: Riluzole in Huntington's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIL_DE1_201
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Riluzole

SUMMARY:
Primary objective:

* The primary objective of the study is to establish that riluzole slows down (1) the decrease in total functional capacity (TFC), (2) the increase of the motor score of the Unified Huntington's Disease Rating Scale (UHDRS) as well as (3) the increase of a combined score of these.

Secondary objectives:

Secondary objectives are to assess

* changes in the other UHDRS subscales
* the number of patients who need antichoreic treatment and the time until this treatment has to be initiated
* the safety/tolerability of riluzole in Huntington patients

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Huntington's disease and CAG repeat length of 36 or more
* UHDRS Motor score of at least 5 points
* UHDRS TFC score of at least 8 points, i.e. patients must be independently ambulatory and must not require nursing care
* Females require a negative blood pregnancy test at inclusion

Exclusion Criteria:

* Any forms of chorea other than Huntington's disease
* Patients on antichoreic treatment within one month prior to entry or foreseen to require such treatment within the first 3 months after randomization (antichoreic medication is prohibited during entire study)
* Other unacceptable prior/concomitant medications
* Uncontrolled major psychiatric disorders, in particular uncontrolled major depression (DSM IV definition)
* Drug or alcohol dependence and/or abuse (DSM IV definition) within the past 6 months
* Any other concomitant disease with a reasonable possibility to interfere with the study
* Females who are breast-feeding, not sterilized, at least one year postmenopausal or don't use an adequate contraceptive method for at least one month prior to and during study participation
* Participation in another clinical study with any investigational drug within 30 days prior to study screening
* Prior exposure to riluzole
* ALT and/or AST and/or Total Bilirubin levels greater than 1.5 times the upper limits of normal range, or hepatic disease other than Gilbert's disease
* Creatinine serum concentrations above 200 µmol/l (resp. 2,3 mg/dl) or hematology parameters as follows: Hemoglobin smaller 11 g/dl for males resp. smaller 10 g/dl for females, or White Blood Cell smaller 3,5 x 10000000000/l

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 1999-11; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
UHDRS-motor score, TFC

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

REFERENCES:
- [Derived] Schramm C, Katsahian S, Youssov K, Demonet JF, Krystkowiak P, Supiot F, Verny C, Cleret de Langavant L, Bachoud-Levi AC; European Huntington's Disease Initiative Study Group and the Multicentre Intracerebral Grafting in Huntington's Disease Group. How to Capitalize on the Retest Effect in Future Trials on Huntington's Disease. PLoS One. 2015 Dec 29;10(12):e0145842. doi: 10.1371/journal.pone.0145842. eCollection 2015. PMID 26714284